CLINICAL TRIAL: NCT00767013
Title: Preoperative Assessment of Aortic Valve Stenosis and Coronary Artery Disease: Dual-source Computed Tomography Compared With Invasive Coronary Angiography and Transthoracic Echocardiography
Brief Title: Preoperative Assessment of Aortic Valve Stenosis and Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Luzerner Kantonsspital (Other)
Responsible Party: Principal Investigator, Prof. Paul Erne, Prof. Paul Erne, Luzerner Kantonsspital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cardiac imaging DSCT
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Aortic Valve Stenosis; Coronary Disease
Keywords: DSCT, coronary artery disease, aortic valve stenosis
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Disease; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AVS, CAD (Experimental): DSCT
  Interventions: Other: DSCT, TTE

INTERVENTIONS:
Other: DSCT, TTE — One assessment each

SUMMARY:
We sought to determine whether the dual-source computed tomography assessment of aortic valve stenosis and coronary artery disease is equivalent to or even better than conventional invasive coronary angiography and transthoracic echocardiography.

DETAILED DESCRIPTION:
Until now invasive coronary angiography has established itself for the assessment of symptomatic aortic valve stenosis. Literature shows a good correlation between MSCT, MRI, TTE and TEE for evaluating the severity of the aortic valve stenosis.

The dual-source computed tomography (DSCT) is capable of assessing coronary arteries with a high sensitivity and specificity in term of relevant stenosis (>50%), due to its excellent spatial and temporal resolution. This study includes the assessment of patients with symptomatic valve stenosis. The severity of the aortic valve stenosis is being assessed by DSCT and TTE. Significant coronary artery stenosis and its localisation are assessed by DSCT and invasive coronary angiography. We examine the correlation between DSCT on one side and either TTE or invasive coronary angiography on the other.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aortic valve disease who were scheduled to undergo cardiac surgery

Exclusion Criteria:

* Hemodynamic instability
* Renal insufficiency (serum creatinine level > 133umol/L)
* Known allergy to iodinated contrast agents
* Non-treated hyperthyreosis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2007-05; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Quality of cardiac imaging in computed tomography | After comparison of imaging measurements

CONTACTS AND LOCATIONS:
Overall Officials: Paul Erne, MD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Department of Cardiology, Lucerne, Canton of Lucerne, Switzerland